CLINICAL TRIAL: NCT04024904
Title: Virtual Reality Hypnosis Distraction Utility to Improve the Quality of Routine Procedure-related Pain During Preoperative Locoregional Anaesthesia
Brief Title: Virtual Reality Hypnosis Distraction Utility to Improve Tolerance to Regional Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Van Hecke Delphine, Principal Investigator, attending physician, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B406201836302
Record Dates: First submitted 2019-04-18; First posted 2019-07-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia
Keywords: regional anesthesia; virtual reality; hypnosis; distraction

STUDY DESIGN:
Intervention Model Description: The Virtual Hypnosis Reality Distraction (VHRD) technique is the program of OncomfortTM (Oncomfort Inc, Houston, USA). The OncomfortTM device include the hyper vision 3D virtual reality glasses and disposable single-patient-use headphones. The program is an immersive experience focused on inducing relaxation environment and this program exist in 5,15 and 30 minutes.
  In the group VHRD 1 and 2 we use the program throughout the regional block. The time choose for the VHRD program is 15 or 30 min depending of the time required for the regional procedure.
  In the group VHRD 2, we use the program of 5 min and we applied the device before the regional procedure.
Who Masked: Outcomes Assessor
Masking Description: Patients were coached by a separate practitioner aside from the regional anaesthesiologist performing the regional block. The anesthetists in charge of the patient were not blinded, but data collection and statistical analysis were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (No Intervention): In the control group, the patient received the standard pharmacologic intravenous sedation before the regional anaesthesia (2 mg midazolam + 5 µg de sufentanil) without VRHD (Virtual Reality Hypnosis Distraction).
- VRHD1 (Experimental): In the study group VRHD (Virtual Reality Hypnosis Distraction) 1, the patient received the VHRD technique during the peripheral nerve block and received a pharmacologic intravenous sedation only if the patient's asked for it or if the patient shows some discomfort (behavioural pain scale score >3).
  Interventions: Device: OncomfortTM device
- VRHD2 (Experimental): In the study group VRHD (Virtual Reality Hypnosis Distraction) 2, the patient received the VHRD technique for the first time before the regional procedure and a second time during the peripheral nerve block. The patient received a pharmacologic intravenous sedation only if the patient's asked for it or if the patient shows some discomfort (behavioural pain scale score >3).
  Interventions: Device: OncomfortTM device

INTERVENTIONS:
Device: OncomfortTM device — The VHRD (Virtual Reality Hypnosis Distraction) technique is the program of OncomfortTM (Oncomfort Inc, Houston, USA). The OncomfortTM device include the hyper vision 3D virtual reality glasses and disposable single-patient-use headphones. The program is an immersive experience focused on inducing relaxation environment and this program exist in 5,15 and 30 minutes
  Arms: VRHD1; VRHD2

SUMMARY:
Regional anaesthesia has many advantages but it might be a stressful and painful experience. Usually, the anesthetist administers a pharmacologic intravenous sedation to achieve patient's comfort. Though, these medications are not benign, and disadvantages include unpredictable response, adverse effects, and interference with cooperation. The virtual reality hypnosis distraction (VRHD) could be a good non-pharmacological technique to improve patient's comfort, decrease anxiety and procedure related pain. This study is a prospective study where sixty patients scheduled for orthopedic surgery requiring regional anesthesia were randomized in three groups according to the use or not of VRHD during the regional procedure or before as a complementary premedication. The anesthetic management during the regional procedure and the surgery remained otherwise standard for each patient. The first endpoint is the proportion of patients receiving pharmacological sedation (in the VRHD groups compared to the pharmacological sedation group). .

The second endpoint is to determine if the VRHD increases the patient's satisfaction of their anaesthetic management.

The third endpoint is to study various parameters of use of this specific anaesthetic management: time required for the installation and operation time of the VRHD device; the variation of haemodynamic parameters between the separate groups; pain procedure-related and behavioural pain scale scores between the separate groups.

DETAILED DESCRIPTION:
Background Regional anesthesia has many advantages but it might be a stressful and painful experience and the anaesthetist has to establish all the necessary measures to maintain patient's comfort and cooperation. In practice, this ideal situation may be the most challenging part of the regional anesthetic practice. Usually, the anesthetist administers a pharmacologic intravenous sedation, including opioids and benzodiazepines to achieve patient's comfort. These medications are not benign, and disadvantages include possible unpredictable response, adverse effects, and hindered cooperation.

Among the non-pharmacologic techniques which may be used to improve the patient's comfort, decrease anxiety and procedure related pain, hypnosis and virtual reality distraction are increasingly used.

In spite of the encouraging scientific and clinical findings, hypnosis for analgesia is not universally used in medical centers. Its widespread use has been limited by factors such as the advanced expertise, time and effort required by clinicians to provide hypnosis, and the commitment required by patients to engage in hypnosis. It is a challenge to make hypnosis a standard part of care in this environment.

Improvements in technologies made virtual reality (VR) distraction a unique practical tool to provide an immersive, multisensory and three-dimensional (3D) environment that creates a sense of presence which enables to modify the perception of reality and to capture a greater degree of attention. Several theories have been proposed to explain how distraction may inhibit or decrease perception of pain by capturing a greater degree of attention. The "virtual reality analgesia" (= analgesia produces by virtual reality) is a product of the attentional distraction. Hoffmann et al. explained that there is a limit to the conscious attentional resources humans have available to process large amounts of incoming information. Conscious attention is required for pain perception. Hoffmann et al. theorize that the more immersive the VR system, the more attention will be drawn into the virtual world, leaving less attention available to process nociceptive signals.

Until now, VR shows an interest in numerous clinical applications (to help treat anxiety disorders, control pain, support physical rehabilitation, and distract patients during wound care) VR technology guides the patient through the same steps used when hypnosis is induced through an interpersonal process. With attentional mechanisms as a common denominator, the attention-captivating qualities of virtual reality and the suggestion inherent in hypnosis, the potential for a synergistic effect between these modalities is signiﬁcant.

Using a device which combined the advantage of VR technology and hypnosis could probably improve the patient's comfort, decrease his anxiety and procedure related pain.

The first endpoint consist in a significant minimal decrease of 50% of the requirement of IVS delivered to the patient throughout the regional performance, in comparison to the IVS group when using VRHD.

The second endpoint is to determine if VRHD increases patient's satisfaction concerning their anaesthetic management.

The third endpoint is to study various parameters of this specific anesthetic management: time required for the installation and operation time of the VRHD device; variation of haemodynamic parameters; pain procedure-related and behavioural pain scale scores.

Methods Our study is a prospective randomized study. The protocol was approved by the Independent Ethics Committee from Erasmus Hospital.

Written Informed consent was obtained from all participating subjects. Subjects were randomized by the use of a computer-generated random table. Sixty patients scheduled for orthopaedic surgery needing regional anaesthesia are randomized according to the used of VRHD during the regional procedure or before as a complementary premedication.

The patients and the anesthetist in charge of the patient were not blinded but the data collection and statistical analysis were blinded.

Anesthesia management The anesthetic management was standardized for each patient. All subjects were fasting from midnight and premedicated with 0,25-0,5 mg alprazolam per os one hour before the procedure.

During the regional block, the surgical asepsis was respected and the regional block was performed under ultrasound guidance (machine Epic or Philips…). A basic monitoring was installed (EKG (electrocardiogram), NIBP (non-invasive blood pressure), SpO2 (pulse oximetry saturation). A 18 gauge catheter was placed in a vein. To avoid hypoxemia, all patients benefited of a supplemental nasal oxygen (3l/min) if the SpO2 < 95%.

Intraoperatively, the patient was maintained under sedation or general anesthesia according to the surgical prerequisites.

In the postoperative period, standard care was provided to the patient at the postoperative care unit according the American society of anesthesiologists (ASA) recommendations.

Study protocol In the control group, the patient received the standard pharmacologic intravenous sedation before the regional anaesthesia (2 mg midazolam + 5 µg de sufentanil) without VRHD.

In the study group VRHD 1, the patient received the VHRD technique during the peripheral nerve block and received a pharmacologic intravenous sedation only if the patient's asked for it or if the patient shows some discomfort (behavioural pain scale score >3).

In the study group VRHD 2, the patient received the VHRD technique a first time before the regional procedure and a second time during the peripheral nerve block. The patient received a pharmacologic intravenous sedation only if the patient's asked for it or if the patient shows some discomfort (behavioural pain scale score >3).

Virtual reality hypnosis distraction protocol The VHRD technique is the program of OncomfortTM (Oncomfort Inc, Houston, USA). The OncomfortTM device include the hyper vision 3D virtual reality glasses and disposable single-patient-use headphones. The program is an immersive experience focused on inducing relaxation environment and this program exists in durations of 5,15 and 30 minutes.

In the group VHRD 1 and 2, the investigators use the program throughout the regional block. The duration chosen for the VHRD program was 15 or 30 min depending of the time required for the regional procedure.

In the group VHRD 2, the investigators use the program of 5 min for the session occuring before the regional procedure, followed by a 15 or 30 min program during the regional procedure.

Patients were coached by a separate practitioner aside from the regional anesthesiologist performing the regional block.

Study Outcomes The first endpoint consist in a significant minimal decrease of 50% of the requirement of IVS (opioids (µg) and benzodiazepine (mg)) delivered to the patient throughout the regional performance, in comparison to the IVS group when using VRHD.

The second endpoint is to determine if the VRHD increases the patient's satisfaction of their anaesthetic management.

The third endpoint is to study various parameters of this specific anesthetic management: time required for the use and installation of the VRHD device; variation of hemodynamic parameters between the separate groups, pain procedure-related and behavioural pain scale scores between the separate groups;

Statistical Analysis As the first endpoint is to determine if the VRHD decreases the need of pharmacologic intravenous sedation of 50%, the sample size (N=60) is determined by an intention-to-treat test (control group n=20, VRHD 1 n= 20 and VRHD n= 20).

ELIGIBILITY:
Inclusion Criteria:

undergoing elective orthopedic surgery with regional anaesthesia (peripheral nerve block), were aged ≥ 18 years

Exclusion Criteria:

ASA (American Society of anesthesiologists) IV, spinal anesthesia, claustrophobia, blindness, deafness, unable to complete a satisfaction survey, previously documented history of neurologic disease, lack of written informed consent, urgent surgery, allergy to a drug used within the study, ongoing pregnancy, patient's infectious isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving pharmacological sedation | immediately after the regional procedure
  Collecting the proportion of patients (n) receiving pharmacological sedation as opioids (micrograms) and benzodiazepine (milligrams) from the beginning to the end of the regional procedure.

SECONDARY OUTCOMES:
patient's satisfaction with visual analogue scale(VAS) (a range of scores from 0-10) | immediately after regional procedure
  The patient's satisfaction score is determined by measuring the distance (cm) on the 10 cm line between the "no satisfaction" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater satisfaction. Based on the distribution of satisfaction VAS scores during the regional procedure who described their satisfaction as none, moderate or very good, the following cut points on the satisfaction VAS have been decided: no satisfaction (0-4cm), moderate satisfaction (4,1-7 cm), and very satisfaction (7,1-10 cm).

OTHER OUTCOMES:
placement of the VRHD (virtual Reality Hypnosis Distraction) device | once, before the regional procedure
  Collecting the time required for the used or placement of the VRHD (virtual Reality Hypnosis Distraction) device (minutes) before the regional procedure.
heart rate before (bpm) | once, before the regional procedure
  Collecting the patient's heart rate (bpm) before the regional procedure
heart rate after (bpm) | immediately after the regional procedure
  Collecting the patient's heart rate (bpm) after the regional procedure
blood pressure before (mmHg) | once, before the regional procedure
  Collecting the patient's blood pressure (mmHg) before the regional procedure.
blood pressure before (mmHg) | immediately after the regional procedure
  Collecting the patient's blood pressure (mmHg) after the regional procedure.
Patient's comfort score with visual analogue scale (VAS) (a range of scores from 0-10) | immediately after the regional procedure
  The patient's comfort score is determined by measuring the distance (cm) on the 10 cm line between the "no comfort" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater comfort. Based on the distribution of comfort VAS scores during the regional procedure who described their comfort as none, moderate or very good, the following cut points on the comfort VAS have been decided: no comfort (0-4cm), moderate comfort (4,1-7 cm), and very good (7,1-10 cm).

CONTACTS AND LOCATIONS:
Locations (1):
- ULB-Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hu P, Harmon D, Frizelle H. Patient comfort during regional anesthesia. J Clin Anesth. 2007 Feb;19(1):67-74. doi: 10.1016/j.jclinane.2006.02.016. PMID 17321932
- [Result] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Result] Pandya PG, Kim TE, Howard SK, Stary E, Leng JC, Hunter OO, Mariano ER. Virtual reality distraction decreases routine intravenous sedation and procedure-related pain during preoperative adductor canal catheter insertion: a retrospective study. Korean J Anesthesiol. 2017 Aug;70(4):439-445. doi: 10.4097/kjae.2017.70.4.439. Epub 2017 Mar 15. PMID 28794840
- [Result] Mulier JP. Perioperative opioids aggravate obstructive breathing in sleep apnea syndrome: mechanisms and alternative anesthesia strategies. Curr Opin Anaesthesiol. 2016 Feb;29(1):129-33. doi: 10.1097/ACO.0000000000000281. PMID 26595546
- [Result] Guenther U, Riedel L, Radtke FM. Patients prone for postoperative delirium: preoperative assessment, perioperative prophylaxis, postoperative treatment. Curr Opin Anaesthesiol. 2016 Jun;29(3):384-90. doi: 10.1097/ACO.0000000000000327. PMID 26905874
- [Result] Wobst AH. Hypnosis and surgery: past, present, and future. Anesth Analg. 2007 May;104(5):1199-208. doi: 10.1213/01.ane.0000260616.49050.6d. PMID 17456675
- [Result] Hauser W, Hagl M, Schmierer A, Hansen E. The Efficacy, Safety and Applications of Medical Hypnosis. Dtsch Arztebl Int. 2016 Apr 29;113(17):289-96. doi: 10.3238/arztebl.2016.0289. PMID 27173407
- [Result] Askay SW, Patterson DR, Sharar SR. VIRTUAL REALITY HYPNOSIS. Contemp Hypn. 2009 Mar;26(1):40-47. doi: 10.1002/ch.371. PMID 20737029
- [Result] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Result] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Result] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Result] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Result] Carrougher GJ, Hoffman HG, Nakamura D, Lezotte D, Soltani M, Leahy L, Engrav LH, Patterson DR. The effect of virtual reality on pain and range of motion in adults with burn injuries. J Burn Care Res. 2009 Sep-Oct;30(5):785-91. doi: 10.1097/BCR.0b013e3181b485d3. PMID 19692911
- [Result] Furman E, Jasinevicius TR, Bissada NF, Victoroff KZ, Skillicorn R, Buchner M. Virtual reality distraction for pain control during periodontal scaling and root planing procedures. J Am Dent Assoc. 2009 Dec;140(12):1508-16. doi: 10.14219/jada.archive.2009.0102. PMID 19955069
- [Result] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Result] Hoffman HG, Garcia-Palacios A, Patterson DR, Jensen M, Furness T 3rd, Ammons WF Jr. The effectiveness of virtual reality for dental pain control: a case study. Cyberpsychol Behav. 2001 Aug;4(4):527-35. doi: 10.1089/109493101750527088. PMID 11708732
- [Result] Morris LD, Louw QA, Crous LC. Feasibility and potential effect of a low-cost virtual reality system on reducing pain and anxiety in adult burn injury patients during physiotherapy in a developing country. Burns. 2010 Aug;36(5):659-64. doi: 10.1016/j.burns.2009.09.005. Epub 2009 Dec 21. PMID 20022431